CLINICAL TRIAL: NCT05552456
Title: Mid Upper Arm Circumference Versus International Screening Questionnaires in Evaluation of Nutritional Status of Children Attending Assiut University Hospital.
Brief Title: Mid Upper Arm Circumference in Evaluation of Nutrition
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aghapy Gamal Zahy Shafik (Other)
Responsible Party: Sponsor-Investigator, Aghapy Gamal Zahy Shafik, Resident doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Mid upper arm circumference
Record Dates: First submitted 2022-09-19; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assess validity of MUAC versus international screening questionnaires in evaluation of nutritional status of infants and children attending Assiut university children hospital.

DETAILED DESCRIPTION:
Identification of children at risk of malnutrition is essential in treating disease-related malnutrition and optimising the health of all hospitalised patients. Malnutrition is: "the state of nutrition in which a deficiency or excess or imbalance) of energy, protein,and other nutrients causes measurable adverse effects on tissue/body function and clinical outcome"( Elia M et al; 2005)

Mid-upper arm circumference (MUAC) is an alternate nutritional measure that can be used as a possible predictor of weight-for -height irrespective of age. MUAC measurement is a simple, non-invasive, rapid and inexpensive tool for screening malnutrition. Therefore, World Health Organization (WHO) has suggested for evaluation of MUAC for screening at the community level.(Geneva et al; 2020)

Subjective Global Assessment (SGA), a method of nutritional assessment based on clinical judgment, has been widely used to assess the nutritional status for both clinical and research purposes.( Am J Clin Nutr et al; 2007) Because nutritional assessment is difficult, a new technique called Subjective Global Assessment (SGA) was developed. Its ratings have been found to be highly predictive of outcome.4 The procedure is easy to learn and simple to implement. SGA requires no additional laboratory testing or capital outlay. In addition, SGA has been found to correlate strongly with other subjective and objective measures of nutrition( Covinsky KE et al; 2004)

SGA classifies the patient as:

A. Well-nourished B. Mildly malnourished or suspected of malnutrition C. Severely malnourished Clinicians place the patient into one of these categories based upon their subjective rating of the patient in two broad areas: 1. Medical History, 2. Physical Examination.

In general, 60% of the clinician's rating of the patient is based on the results of the medical history, and 40% on the physical examination(see SGA evaluation form)( Covinsky KE et al; 2004)

Medical History Section

The first SGA component, the medical history, involves asking questions and evaluating the patient's answers about the following four parameters:

1. Weight change
2. Dietary intake
3. Gastrointestinal symptoms
4. Functional impairment The patient is rated as either nourished, mildly, moderately malnourished, or severely malnourished for each of the four parameters.

Physical Examination Section Physical evidence of malnutrition is rated differently. There are four categories to select from: normal nutrition, mild malnutrition, moderate malnutrition, or severe malnutrition.

Physical signs to examine include:

1. Loss of subcutaneous fat
2. Muscle wasting
3. Edema
4. Ascites (in hemodialysis patients only) There are several body locations to examine for each parameter(Covinsky KE et al; 2004)

Anthropometric measurments: Anthropometry is the most used tool for nutitional assessment, since it is non-invasive, cheap and it presents quite satisfactory results. In the anthropometric assessment of children's nutritional status, the variables weight, height (or lengh), sex, and age are comined to form anthropometric indices. These are currently expressed as persentiles or z-scores units. The values obtained in the assassed subjects are compared with those produced from a healthy population,which constitute the anthropometric standards (Da Silva et al; 2020)

Screening Tools For Assessment of Malnutrition in Pediatrics(STAMP) : STAMP is nutrition screening tool widely used in children. It considers the present state of medical condition, nutritional intake and history of weight changes. It was published in 2012 after the pilot study among hospitalized children in the UK. It has also been validated in developed and developing countries(Ong SH et al; 2019)

Screening Tool for Risk on Nutritinal Status and Growth (STRONG): STRONG kids developed for hospitalized children. This nutritional risk-screening questionnaire consists of four items: high-risk disease, subjective clinical assessment, nutritional intake and losses, and weight loss or poor weight gain, and each item is allocated a score of 1or 2 points with a maximum total score of 5 points Questions answered unclear were classified as no. A child with a STRONG kids risk score of 0,1-3, or 4-5 has, respectively, a lowm moderate, or high risk of developing malnutrition(Joosten K et al; 2016)

Paediatric Yorkhill Malnutrition Score (The PYMS): form is presented as a simple structured questionnaire, consisting of four questions (steps) which are strong predictors/symptoms of malnutrition. Each of these steps bears a score from 0 to 2 and an overall nutritional risk score (step 5) is calculated based on the sum of the results of steps 1 action plan follows outlined below:

Step 1: Body Mass Index (BMI) STEP 2: Recent Weight Loss STEP 3: Assess Recent Change in Diet/Nutritional Support (for at least the last week) STEP 4: Acute Admission/Condition Effect on Nutrition (at least the next week) STEP 5: Total Nutrition Risk Score and Action Plan( NHS Greater Glasgow and Clyde et al; 2009)

ELIGIBILITY:
Inclusion Criteria:

1. Children aged from 6 months up to 5 years.
2. Both sexes are included

Exclusion Criteria:

- 1-Any children with congenital anomalies. 2-Children diagnosd with genetic diseases. 3-Children with chronic illness. 4-Children younger than 6 months or older than 5 years. 5-Any children whose parents refuse participating in the study.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Descriptve cross sectional study that will be conducted on 500 infants and children to assess the validity of MUAC versus international screening questionnaires in evaluation of nutritional status of those infants and children.
Sampling Method: Non-Probability Sample
Enrollment: 537 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Assess validity of MUAC versus international screening questionnaires in evaluation of nutritional status of infants and children attending Assiut university children hospital. | One year
  Identify value of nutritional screening tools and anthropometric measurements in evaluation of nutritional status of children and to determine which of them has the highest accuracy to be used in daily practice

CONTACTS AND LOCATIONS:
Overall Officials: Osama Mahmoud Elasheer, Study Director — Professor of pediatrics; Amir Mohammed Abo-elgheet, Study Chair — Assistant professor

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elia M, Ljungqvist O and Dowsett J (2005) Principal of Clinical Nutrition:Contrasting the Practice of Nutrition in Health and Disease. Oxford, Blackwell Science Ltd
- [Background] Guideline: Updates on the Management of Severe Acute Malnutrition in Infants and Children. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK190328/ PMID 24649519
- [Background] Secker DJ, Jeejeebhoy KN. Subjective Global Nutritional Assessment for children. Am J Clin Nutr. 2007 Apr;85(4):1083-9. doi: 10.1093/ajcn/85.4.1083. PMID 17413109
- [Background] Covinsky KE, Martin GE, Beyth RJ, Justice AC, Sehgal AR, Landefeld CS. The relationship between clinical assessments of nutritional status and adverse outcomes in older hospitalized medical patients. J Am Geriatr Soc. 1999 May;47(5):532-8. doi: 10.1111/j.1532-5415.1999.tb02566.x. PMID 10323645
- [Background] Ferreira HDS. Anthropometric assessment of children's nutritional status: a new approach based on an adaptation of Waterlow's classification. BMC Pediatr. 2020 Feb 11;20(1):65. doi: 10.1186/s12887-020-1940-6. PMID 32046666
- [Background] Ong SH, Chee WSS, Lapchmanan LM, Ong SN, Lua ZC, Yeo JX. Validation of the Subjective Global Nutrition Assessment (SGNA) and Screening Tool for the Assessment of Malnutrition in Paediatrics (STAMP) to Identify Malnutrition in Hospitalized Malaysian Children. J Trop Pediatr. 2019 Feb 1;65(1):39-45. doi: 10.1093/tropej/fmy009. PMID 29514329
- [Background] Joosten K, van der Velde K, Joosten P, Rutten H, Hulst J, Dulfer K. Association between nutritional status and subjective health status in chronically ill children attending special schools. Qual Life Res. 2016 Apr;25(4):969-77. doi: 10.1007/s11136-015-1130-4. Epub 2015 Sep 11. PMID 26362418
- [Background] Nutrition Tool Steering Group, Women and children's Directorate, NHS Greater Glasgow and Clyde, 2009.